CLINICAL TRIAL: NCT01874002
Title: Multicenter, Prospective, Clinical Outcomes After Deployment of the Abluminal Sirolimus Coated Bio-Engineered Stent (Combo Bio- Engineered Sirolimus Eluting Stent) Post Market Registry
Brief Title: Prospective Registry to Asses the Long-term Safety and Performance of the Combo Stent
Acronym: REMEDEE Reg
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Robbert J de Winter (Other)
Responsible Party: Sponsor-Investigator, Robbert J de Winter, Professor of Clinical Cardiology, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: W12_186; Version 2.0 (Registry Identifier: RoPR ID: 102)
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease
Keywords: Stents; Stent; Drug eluting; Drug eluting stent; Drug eluting stents; Endothelial progenitor cell; Endothelial progenitor cell capturing; Sirolimus; Sirolimus eluting; Percutaneous Coronary Intervention; PCI; Registry; Registries; Multi center; Multi centre
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Combo stent: Consecutive patients in whom a treatment with a Combo stent in the setting of routine clinical care is attempted are entered into the registry.
  Interventions: Device: Combo stent

INTERVENTIONS:
Device: Combo stent — Percutaneous coronary intervention of patients with an indication for stent treatment with the COMBO stent, a stent with an endothelial progenitor cell attracting coating and abluminal sirolimus matrix. All consecutive patients treated with, or attempted treatment with, a COMBO stent are followed by telephone contact for 5 years.
  Other Names: Abluminal Sirolimus Coated Bio-Engineered Stent; Combo Bio-Engineered Sirolimus Eluting Stent; SirolimusECS

SUMMARY:
Patients with stenosis in one or more coronary artery are often treated with a percutaneous coronary intervention (PCI). As part of the PCI treatment a stent is often placed to keep the vessel open over time.

The Combo-Stent is a novel stent for use during percutaneous angioplasty. In short, the Combo stent combines a drug eluting technique and an endothelial cell attracting layer. The drug coating is designed to prevent re-narrowing of the stent. The endothelial cell attracting layer is designed to ensure rapid coverage of the stent struts with vascular wall cells.

The REMEDEE REGISTRY evaluates the long-term safety and performance of the Combo stent in routine clinical practice. In total 1000 patients will be registered and followed for five years.

DETAILED DESCRIPTION:
Registry Investigated Device:

The OrbusNeich Combo Bio-engineered Sirolimus Eluting Stent (Combo Stent) consists of a 316L stainless steel alloy abluminally coated with a biocompatible, biodegradable polymer containing sirolimus. Covalently attached to this matrix is a layer of murine, monoclonal, anti-human CD34 antibody. The antibody specifically targets CD34+ cells in circulation. Endothelial progenitor cells (EPCs) are CD34+. The stent is supplied premounted on a 0.014" guide wire compatible low profile rapid exchange balloon catheter delivery system. The Combo Stent is Conformitée Européenne (CE) marked.

Registry Objectives:

The REMEDEE REGISTRY evaluates the long term safety and performance of the Abluminal Sirolimus Coated Bio-Engineered Stent (Combo Bio-Engineered Sirolimus Eluting Stent) in routine clinical practice. The primary objective of the registry is to evaluate the one year incidence of target lesion failure in consecutive patients undergoing percutaneous coronary intervention with (attempted) Combo stent placement.

Registry Design:

The REMEDEE REGISTRY is an international, prospective, multicenter, cohort post market registry with five years follow-up to evaluate outcomes in patients undergoing percutaneous coronary intervention with (attempted) Combo stent placement. The registry population consists of consecutive patients in whom a treatment with a Combo stent in the setting of routine clinical care is attempted.

This registry involves the collection of baseline demographic, clinical, and angiographic data, as well as follow-up data in consecutive patients in whom the Combo stent is used to treat (a) coronary lesion(s) in the setting of routine clinical care. Patients are registered in up to 10 European high volume PCI centers. A follow-up is scheduled at 30 days, 180 days,1 year, 2 years, 3 years, 4 years and 5 years post procedure. Follow-up is obtained at a planned regular visit to the out-patient clinic, or by telephone contact with the patient.

Quality control:

All data will be entered on-site in an electronic case report (eCRF) form according to Good Clinical Practice guidelines.

All sites will monitored regularly during the time of the registry. The monitor plan involves a hundred percent procedural information and event monitoring. During data monitoring, all source data will be assessed for accuracy, completeness, and representativeness of registry data by comparing the data to external data sources. Data checks to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry are implemented in the (eCRF). A data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, coding information if used, and normal ranges if relevant is part of the database and eCRF design. Standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management are in place. A detailed statistical analysis plan describing the analytical principles and statistical techniques to be employed in order to address the primary and secondary objectives, as specified in the study protocol is available. Missing data is accounted for in the design of the eCRF template, and will be handled according to the statistical plan.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients eligible for Combo stent placement by percutaneous coronary intervention are included in the REMEDEE REGISTRY

Exclusion Criteria:

* High probability of non-adherence to the follow-up requirements (due to social, psychological or medical reasons)
* Currently participating in another investigational drug or device study in which a routine angiographic follow-up is planned
* A life expectancy of <1 year
* Explicit refusal of participation in the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry population consists of consecutive patients in whom a treatment with a Combo stent in the setting of routine clinical care is attempted.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Adjudicated Target Lesion Failure | 1 year post-procedure
  Adjudicated device-oriented composite target lesion failure (TLF) defined as a composite of cardiac death, non-fatal myocardial infarction (MI) not clearly attributable to a nontarget vessel, or target lesion revascularization (TLR) (percutaneous or by coronary artery bypass grafting).

SECONDARY OUTCOMES:
Adjudicated Target Lesion Failure | 30 days post-procedure
  Adjudicated device-oriented composite target lesion failure (TLF) defined as a composite of cardiac death, non-fatal myocardial infarction (MI) not clearly attributable to a nontarget vessel, or target lesion revascularization (TLR) (percutaneous or by coronary artery bypass grafting).
Adjudicated Target Lesion Failure | 180 days post procedure
  Adjudicated device-oriented composite target lesion failure (TLF) defined as a composite of cardiac death, non-fatal myocardial infarction (MI) not clearly attributable to a nontarget vessel, or target lesion revascularization (TLR) (percutaneous or by coronary artery bypass grafting).
Individual components of target lesion failure (TLF) | 1 year post-procedure
  Individual components of target lesion failure (TLF):
  * Cardiac death
  * Non-fatal MI not clearly attributable to a non-target vessel
  * Target lesion revascularization (TLR)
Individual components of target lesion failure (TLF) | 30 days post-procedure
  Individual components of TLF:
  * Cardiac death
  * Non-fatal MI not clearly attributable to a non-target vessel
  * Target lesion revascularization (TLR)
Individual components of target lesion failure (TLF) | 180 days post-procedure
  Individual components of TLF:
  * Cardiac death
  * Non-fatal MI not clearly attributable to a non-target vessel
  * Target lesion revascularization (TLR)
Individual components of target lesion failure (TLF) | 1 year post-procedure
  Individual components of TLF:
  * Cardiac death
  * Non-fatal MI not clearly attributable to a non-target vessel
  * Target lesion revascularization (TLR)
Adjudicated patient-oriented composite Major Adverse Cardiac Events (MACE) | 1 year post-procedure
  Adjudicated patient-oriented composite MACE as a composite of:
  * All death
  * Any myocardial infarction
  * Any revascularization
Adjudicated patient-oriented composite Major Adverse Cardiac Events (MACE) | 30 days post-procedure
  Adjudicated patient-oriented composite MACE as a composite of:
  * All death
  * Any myocardial infarction
  * Any revascularization
Adjudicated patient-oriented composite Major Adverse Cardiac Events (MACE) | 180 days post-procedure
  Adjudicated patient-oriented composite MACE as a composite of:
  * All death
  * Any myocardial infarction
  * Any revascularization
Each of the individual components of Major Adverse Cardiac Events(MACE) | 1 year post-procedure
  Each of the individual components of MACE:
  * All death
  * Any myocardial infarction
  * Any revascularization
Adjudicated stent thrombosis (definite/probable/possible) | 1 year post-procedure
  Adjudicated stent thrombosis (definite/probable/possible) per Academic Research Consortium definitions
Adjudicated stent thrombosis (definite/probable/possible) | 30 days post-procedure
  Adjudicated stent thrombosis (definite/probable/possible) per Academic Research Consortium definitions
Adjudicated stent thrombosis (definite/probable/possible) | 180 days post-procedure
  Adjudicated stent thrombosis (definite/probable/possible) per Academic Research Consortium definitions
Device success | Procedural
  Percentage of patients with a successful delivery and deployment of the Combo stent to the target lesion and a final diameter stenosis after stenting ≤20% by visual assessment in the presence of grade 3 TIMI flow, by visual estimation
Procedure success | Procedural
  Successful stent placement and no periprocedural complications.
Adjudicated Target Lesion Failure | 2 years post-procedure
  Adjudicated device-oriented composite target lesion failure (TLF) defined as a composite of cardiac death, non-fatal myocardial infarction (MI) not clearly attributable to a nontarget vessel, or target lesion revascularization (TLR) (percutaneous or by coronary artery bypass grafting).
Adjudicated Target Lesion Failure | 3 years post-procedure
  Adjudicated device-oriented composite target lesion failure (TLF) defined as a composite of cardiac death, non-fatal myocardial infarction (MI) not clearly attributable to a nontarget vessel, or target lesion revascularization (TLR) (percutaneous or by coronary artery bypass grafting).
Adjudicated Target Lesion Failure | 4 years post-procedure
  Adjudicated device-oriented composite target lesion failure (TLF) defined as a composite of cardiac death, non-fatal myocardial infarction (MI) not clearly attributable to a nontarget vessel, or target lesion revascularization (TLR) (percutaneous or by coronary artery bypass grafting).
Adjudicated Target Lesion Failure | 5 years post-procedure
  Adjudicated device-oriented composite target lesion failure (TLF) defined as a composite of cardiac death, non-fatal myocardial infarction (MI) not clearly attributable to a nontarget vessel, or target lesion revascularization (TLR) (percutaneous or by coronary artery bypass grafting).
Individual components of target lesion failure (TLF) | 2 years post-procedure
  Individual components of target lesion failure (TLF):
  * Cardiac death
  * Non-fatal MI not clearly attributable to a non-target vessel
  * Target lesion revascularization (TLR)
Individual components of target lesion failure (TLF) | 3 years post-procedure
  Individual components of target lesion failure (TLF):
  * Cardiac death
  * Non-fatal MI not clearly attributable to a non-target vessel
  * Target lesion revascularization (TLR)
Individual components of target lesion failure (TLF) | 4 years post-procedure
  Individual components of target lesion failure (TLF):
  * Cardiac death
  * Non-fatal MI not clearly attributable to a non-target vessel
  * Target lesion revascularization (TLR)
Individual components of target lesion failure (TLF) | 5 years post-procedure
  Individual components of target lesion failure (TLF):
  * Cardiac death
  * Non-fatal MI not clearly attributable to a non-target vessel
  * Target lesion revascularization (TLR)
Adjudicated patient-oriented composite Major Adverse Cardiac Events (MACE) | 2 years post-procedure
  Adjudicated patient-oriented composite MACE as a composite of:
  * All death
  * Any myocardial infarction
  * Any revascularization
Adjudicated patient-oriented composite Major Adverse Cardiac Events (MACE) | 3 years post-procedure
  Adjudicated patient-oriented composite MACE as a composite of:
  * All death
  * Any myocardial infarction
  * Any revascularization
Adjudicated patient-oriented composite Major Adverse Cardiac Events (MACE) | 4 years post-procedure
  Adjudicated patient-oriented composite MACE as a composite of:
  * All death
  * Any myocardial infarction
  * Any revascularization
Adjudicated patient-oriented composite Major Adverse Cardiac Events (MACE) | 5 years post-procedure
  Adjudicated patient-oriented composite MACE as a composite of:
  * All death
  * Any myocardial infarction
  * Any revascularization
Adjudicated stent thrombosis (definite/probable/possible) | 2 years post-procedure
  Adjudicated stent thrombosis (definite/probable/possible) per Academic Research Consortium definitions
Adjudicated stent thrombosis (definite/probable/possible) | 3 years post-procedure
  Adjudicated stent thrombosis (definite/probable/possible) per Academic Research Consortium definitions
Adjudicated stent thrombosis (definite/probable/possible) | 4 years post-procedure
  Adjudicated stent thrombosis (definite/probable/possible) per Academic Research Consortium definitions
Adjudicated stent thrombosis (definite/probable/possible) | 5 years post-procedure
  Adjudicated stent thrombosis (definite/probable/possible) per Academic Research Consortium definitions

CONTACTS AND LOCATIONS:
Overall Officials: Robbert J de Winter, MD, PhD, Principal Investigator — Academic Medical Centre - University of Amsterdam
Locations (9):
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- Netherlands (5):
  - Academic Medical Center - University of Amsterdam, Amsterdam
  - Ter Gooi Ziekenhuizen, Blaricum
  - Amphia Ziekenhuis, Breda
  - Radboud UMC, Nijmegen
  - Isala Klinieken, Zwolle
- Meixoeiro Hospital, Vigo, Spain
- Craigavon Cardiac Centre, Craigavon, United Kingdom

REFERENCES:
- [Background] Granada JF, Inami S, Aboodi MS, Tellez A, Milewski K, Wallace-Bradley D, Parker S, Rowland S, Nakazawa G, Vorpahl M, Kolodgie FD, Kaluza GL, Leon MB, Virmani R. Development of a novel prohealing stent designed to deliver sirolimus from a biodegradable abluminal matrix. Circ Cardiovasc Interv. 2010 Jun 1;3(3):257-66. doi: 10.1161/CIRCINTERVENTIONS.109.919936. Epub 2010 May 4. PMID 20442358
- [Background] Nakazawa G, Granada JF, Alviar CL, Tellez A, Kaluza GL, Guilhermier MY, Parker S, Rowland SM, Kolodgie FD, Leon MB, Virmani R. Anti-CD34 antibodies immobilized on the surface of sirolimus-eluting stents enhance stent endothelialization. JACC Cardiovasc Interv. 2010 Jan;3(1):68-75. doi: 10.1016/j.jcin.2009.09.015. PMID 20129572
- [Derived] Chandrasekhar J, Kok MM, Kalkman DN, Aquino MB, Zocca P, Woudstra P, Beijk MA, Kerkmeijer LS, Sartori S, Baber U, Tijssen JG, Koch KT, Dangas GD, Colombo A, Pocock S, von Birgelen C, Mehran R, de Winter RJ; COMBO Collaborators and BIO-RESORT Investigators. 1-Year Clinical Outcomes of All Comers Treated With 2 Bioresorbable Polymer-Coated Sirolimus-Eluting Stents: Propensity Score-Matched Comparison of the COMBO and Ultrathin-Strut Orsiro Stents. JACC Cardiovasc Interv. 2020 Apr 13;13(7):820-830. doi: 10.1016/j.jcin.2019.11.023. PMID 32273094
- [Derived] Chandrasekhar J, Kerkmeijer LS, Kalkman DN, Sartori S, Aquino MB, Woudstra P, Beijk MA, Tijssen JG, Koch KT, Hajek P, Atzev B, Hudec M, Ong TK, Mates M, Borisov B, Warda HM, den Heijer P, Wojcik J, Iniguez A, Coufal Z, Khashaba A, Munawar M, Gerber RT, Yan BP, Lee M, Baber U, Dangas GD, Colombo A, de Winter RJ, Mehran R; MASCOT and REMEDEE investigators (full list of collaborators shown in the Appendix). Sex differences in 1-year clinical outcomes after percutaneous coronary intervention with COMBO stents: From the COMBO collaboration. Catheter Cardiovasc Interv. 2021 Apr 1;97(5):797-804. doi: 10.1002/ccd.28853. Epub 2020 Mar 21. PMID 32198837
- [Derived] Kalkman DN, Kerkmeijer LS, Woudstra P, Menown IBA, Suryapranata H, den Heijer P, Iniguez A, van 't Hof AWJ, Erglis A, Arkenbout KE, Muller P, Koch KT, Tijssen JG, Beijk MAM, de Winter RJ. Three-year clinical outcomes after dual-therapy COMBO stent placement: Insights from the REMEDEE registry. Catheter Cardiovasc Interv. 2019 Sep 1;94(3):342-347. doi: 10.1002/ccd.28047. Epub 2018 Dec 18. PMID 30565371
- [Derived] Kalkman DN, Woudstra P, Menown IBA, den Heijer P, Van't Hof AW, Erglis A, Suryapranata H, Arkenbout KE, Iniguez A, Muller P, Tijssen JG, Beijk MAM, de Winter RJ. Two-year clinical outcomes of patients treated with the dual-therapy stent in a 1000 patient all-comers registry. Open Heart. 2017 Jul 11;4(2):e000634. doi: 10.1136/openhrt-2017-000634. eCollection 2017. PMID 28761685
- [Derived] Woudstra P, Kalkman DN, den Heijer P, Menown IB, Erglis A, Suryapranata H, Arkenbout KE, Iniguez A, van 't Hof AW, Muller P, Tijssen JG, de Winter RJ. 1-Year Results of the REMEDEE Registry: Clinical Outcomes After Deployment of the Abluminal Sirolimus-Coated Bioengineered (Combo) Stent in a Multicenter, Prospective All-Comers Registry. JACC Cardiovasc Interv. 2016 Jun 13;9(11):1127-34. doi: 10.1016/j.jcin.2016.02.052. Epub 2016 May 18. PMID 27209254